CLINICAL TRIAL: NCT05547698
Title: Venoarterial ECMO vs Off-Pump Bilateral Orthotopic Lung Transplantation VIP BOLT Trial: A Multicenter Prospective Randomized Trial
Brief Title: A Study of Venoarterial ECMO vs Off-Pump Bilateral Orthotopic Lung Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mauricio A. Villavicencio Theoduloz, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-005691
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Lung Transplant
Keywords: Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Off-Pump Bilateral Lung Transplantation (Active Comparator): Subjects will receive 'off-pump' technique for lung transplantation as part of standard of care
  Interventions: Procedure: Off-pump lung transplantation
- Venoarterial Extra Corporeal Membrane Oxygenation (VA ECMO) Bilateral Lung Transplantation (Active Comparator): Subjects will receive VA ECMO technique for lung transplantation as part of standard of care
  Interventions: Procedure: Venoarterial ECMO lung transplantation

INTERVENTIONS:
Procedure: Off-pump lung transplantation — General anesthesia, intubation with double lumen tube, thoracotomies or clamshell incision, pneumonectomy starting by the less perfused lung in the scan, stump preparation, lung implantation, reperfusion, gradual release of the pulmonary artery clamp, deairing, ventilation of the 1st implanted lung. The process is repeated at the contralateral side. Ventilation of both lungs, chest closure.
  Arms: Off-Pump Bilateral Lung Transplantation
Procedure: Venoarterial ECMO lung transplantation — General anesthesia, intubation with double lumen tube, thoracotomies or clamshell incision, heparin, peripheral or central venoarterial ECMO cannulation, first pneumonectomy, stump preparation, lung implantation, reperfusion, release of the pulmonary artery clamp, deairing, ventilation of the 1st implanted lung. The process is repeated at the contralateral side. Ventilation of both lungs, ECMO decannulation, chest closure.
  Arms: Venoarterial Extra Corporeal Membrane Oxygenation (VA ECMO) Bilateral Lung Transplantation

SUMMARY:
The purpose of this research study is to compare the technique of performing bilateral lung transplantation off-pump vs venoarterial ECMO (VA ECMO). The goal of the trial is to determine which technique has lower rates of primary graft dysfunction.

DETAILED DESCRIPTION:
The Investigators of the Extracorporeal Life Support Registry in Lung Transplantation (ECLS Registry) has studied the impact of the type of intraoperative extracorporeal life support on primary graft dysfunction (PGD) after lung transplantation (LTx) in an international registry. The investigators have demonstrated that severe PGD at 48-72 hours is greater when LTx is performed using cardiopulmonary bypass (CPB) (43%) when compared to veno-arterial (VA) ECMO. However, PGD after VA ECMO remained high (29%) when compared to off-pump (12%). Conversely, there are retrospective series showing that when compared to off-pump technique, VA ECMO has reduced PGD rates and improved survival. Because selection bias and unknown confounders in retrospective studies could have been the cause of these conflicting results, part of the ECLS Registry Investigators are committed to a prospective multicenter randomized trial comparing off-pump versus VA ECMO LTx.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral Lung Transplantation (LTx) recipients.
* Mean pulmonary artery pressure < or = 35 mmHg.
* Eligible for off-pump or VA ECMO based on the judgement of the attending surgeon.

Exclusion Criteria:

* Single lung transplant
* Multiorgan transplant.
* Donor after cardiac death (DCD).
* Re-transplant.
* Intention to use prophylactic post-operative ECMO.
* Previous major lung surgery. Video-assisted thoracoscopic surgery (VATS) and wedge resection are not an exclusion criterion.
* Previous pleurodesis.
* Preoperative ECMO and/or mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-09-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Primary Lung Graft Dysfunction (PGD) grade 3 | 48-72 hours
  Rate of PGD according to the The International Society for Heart and Lung Transplantation (ISHLT) classification
Mortality | 90 days
  Death rate of subjects following lung transplantation
Primary Lung Graft Dysfunction (PGD) grade 3 and Mortality | 48-72 hours and 90 days
  Rate of PGD according to the The International Society for Heart and Lung Transplantation (ISHLT) classification plus the Death rate of subjects following lung transplantation

SECONDARY OUTCOMES:
Red blood cell transfusions | Intraoperative plus the first 24 hours in the ICU
  Number of subjects to require red blood cell transfusions
Chest tube output | First 24 hours
  Chest tube output the first 24 hours following lung transplantation reported in cubic centimeter (cc)
Incidence of re-exploration for bleeding | First 48 hours
  Number of subject to require re-exploration for bleeding
Incidence of air emboli | During VA ECMO run
  Number of subjects to experience air emboli
Incidence of stroke | 90 days or discharge from the index hospitalization
  Number of subjects to experience stroke
Incidence of Primary Lung Graft Dysfunction (PGD) grade 3 | At 0 hours (ICU arrival) and 24 hours
  Number of subjects to experience a PGD grade 3 following lung transplantation. PGD will be rated according to the The International Society for Heart and Lung Transplantation (ISHLT) classification
Incidence of pneumonia | 90 days or discharge from the index hospitalization
  Number of subjects to experience pneumonia
Incidence of need for dialysis | 90 days or discharge from the index hospitalization
  Number of subjects to need dialysis
Incidence of transplant rejection | 90 days or discharge from the index hospitalization
  Number of subjects to experience transplant rejection
Incidence of bronchial dehiscence | 90 days or discharge from the index hospitalization
  Number of subjects to experience bronchial dehiscence
Incidence of tracheostomy | 90 days or discharge from the index hospitalization
  Number of subjects to require tracheostomy
Length of mechanical ventilation | 90 days or discharge from the index hospitalization
  Total amount of time subjects require mechanical ventilation following lung transplantation
Length of stay | 90 days or discharge from the index hospitalization
  Total amount of time subjects are hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Villavicencio, MD, MBA, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - University Of Louisville, Louisville, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials